CLINICAL TRIAL: NCT00585819
Title: Validation of a Novel Thoracic Neoplasm Radiotherapy Image Guidance Technique: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of interest
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HSC-2007-0109
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2. Free breathing (Experimental): Freebreathing in Body fix mold
  Interventions: Procedure: Freebreathing in Body fix mold
- 1. breathing cycle (Experimental): reproducing breathing cycles
  Interventions: Procedure: reproduce breathing cycle utilizing spirometry

INTERVENTIONS:
Procedure: reproduce breathing cycle utilizing spirometry — reproduce breathing cycle utilizing spirometry
  Arms: 1. breathing cycle
Procedure: Freebreathing in Body fix mold — Freebreathing in Body fix mold
  Arms: 2. Free breathing

SUMMARY:
The overall, broad objective of this study is to pilot the BSD technique. The specific purpose of this particular study is to generate pilot data to validate several crucial steps of the BSD technique, in particular steps 1, 2, and 4. Radiation treatments will proceed per standard of care, and will not be modified in any way during this protocol. This study is a non-treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Any thoracic neoplasm scheduled to undergo radiation therapy
* 18 years or older
* Must be treated with radiation as part of standard of care
* Able to tolerate the mouthpiece for spirometry and video glasses
* Ability to provide written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of the guided breathing cycle | 6 weeks

SECONDARY OUTCOMES:
Stability of motion envelope derived from initial 4D imaging compared to CT's obtained throughout the course of therapy | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minesh Mehta, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States